CLINICAL TRIAL: NCT07334444
Title: Current Status Assessment for the Development of a Protocol to Optimize the Management of Obstructive Sleep Apnea (OSA) in Children With Down Syndrome
Brief Title: Optimizing the Management of OSA in Children With Down Syndrome
Acronym: SAOS-21
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9617
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea of Child; Down syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Down Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this retrospective descriptive study is to assess current practices for the screening and surgical treatment of OSA in children with Down syndrome at the Strasbourg University Hospital and to disseminate a management algorithm in France.

ELIGIBILITY:
Inclusion Criteria:

* Child with Down syndrome,
* Aged between 0 and 17 years,
* Having been seen for an ENT consultation at the University Hospital or the Sleep Center of the University Hospital of Strasbourg between January 1, 2019, and December 31, 2024

Exclusion Criteria:

- Presence of a written objection in the medical file of the subject (and/or their representative) to the reuse of their data for scientific research purposes.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: - Child with Down syndrome, aged between 0 and 17 years and having been seen for an ENT consultation at the University Hospital or the Sleep Center of the University Hospital of Strasbourg between January 1, 2019, and December 31, 2024
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) before and after surgery. | Day 1 before surgery and Day 1 after surgery
  The AHI is a number that indicates how many times per hour breathing is abnormal during sleep.
  It adds up:
  * Apneas → breathing stops completely
  * Hypopneas → breathing becomes much shallower
  Scores:
  * AHI < 5 → normal
  * AHI between 5 and 15 → mild impairment
  * AHI between 15 and 30 → moderate impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et de Chirurgie Cervico-faciale - CHU de Strasbourg - France, Strasbourg, France